CLINICAL TRIAL: NCT00345319
Title: Evaluate the Immunogenicity and Safety of Rabies Vaccine Given in a Post-exposure Prophylaxis Regimen to Healthy Children and Adults Aged 10-60 Years.
Brief Title: Purified Rabies Vaccine for Human Use (Chick-embryo Cell)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: M49P7
Record Dates: First submitted 2006-06-27; First posted 2006-06-28 (Estimated); Last update posted 2011-12-14 (Estimated); Status verified 2011-12

CONDITIONS: Rabies Post-exposure Prophylaxis
Keywords: rabies; vaccine; post-exposure prophylaxis
MeSH Terms: conditions — Rabies | interventions — Rabies Vaccines

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Group 1 (Active Comparator)
  Interventions: Biological: rabies vaccine
- Group 2 (Active Comparator)
  Interventions: Biological: rabies vaccine

INTERVENTIONS:
Biological: rabies vaccine — Administration of PCECV according to ESSEN regimen

SUMMARY:
Evaluate the immunogenicity and safety of rabies vaccine given in a post-exposure prophylaxis regimen to healthy children and adults aged 10-60 years.

ELIGIBILITY:
Inclusion Criteria:

* male and female healthy subjects aged 10-60 years old

Exclusion Criteria:

* history of rabies immunization
* previous exposure to a suspect rabid animal within the last 12 months
* any significant acute or chronic infections requiring systemic antibiotic treatment or antiviral therapy within the past 7 days
* treatment with corticosteroids, immunosuppressive or anti-malaria drugs during the two month period before enrollment
* known/suspected immunodeficiency, or autoimmune disease, or any immunologic disorder
* known hypersensitivity to neomycin, tetracycline, amphotericin-B, or any other vaccine component

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 630 (Actual)
Dates: Start 2006-03; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
serum bactericidal activity | measured at day 14 and day 45 after first vaccination dose

SECONDARY OUTCOMES:
solicited local and systemic reactions | within 6 days following vaccination and adverse events thought the study

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines - Information Services, Study Chair — Novartis Vaccines & Diagnostics
Locations (1):
- Danyang CDC, Danyang, Jiangsu, China